CLINICAL TRIAL: NCT04363593
Title: Serology COVID-19 From the Cornwall Hospital Union
Acronym: ROCOCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Cornouaille (Other)
Collaborators: Centre Hospitalier Régional et Universitaire de Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC20.0122
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Corona Virus Infection
Keywords: coronavirus infection; serology
MeSH Terms: conditions — Coronavirus Infections | interventions — Serologic Tests; Serum Bactericidal Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- prospective group COVID (Other): New patients consulting for suspected or diagnosed COVID(+)
  Interventions: Biological: Serological test
- retrospective group COVID (Other): Patients already diagnosed with COVID(+) or with a suspicion of unconfirmed COVID or at a date before the apparition of the COVID infection (April-March 2019)
  Interventions: Biological: Serum test
- Hospital staff (Other): All hospital staff including those already diagnosed at COVID(+)
  Interventions: Biological: Serological test; Biological: Serum test

INTERVENTIONS:
Biological: Serological test — Serological testing is performed for patients with confirmed COVID-19 infection by RT-PCR.
  Arms: Hospital staff; prospective group COVID
Biological: Serum test — Use of the serum taken from patients consulted for suspicion of COVID-19 before the beginning of the trial
  Arms: Hospital staff; retrospective group COVID

SUMMARY:
Coronavirus (COVID-19) is a pandemic-like disease caused by a new coronavirus called Severe Acute Respiratory Syndrome Coronavirus 2 (SARSCoV-2) isolated in China in 2019. Clinical manifestations vary widely from one individual to another, from asymptomatic carrier to a febrile cough that can rapidly lead to acute respiratory distress syndrome. Since the beginning of the COVID-19 epidemic, screening by chest X-ray (RT) and polymerase chain reaction (PCR) SARS-CoV-2 conducted by the Cornwall Hospital Union laboratory has shown that among symptomatic patients and hospital staff suspected of being COVID-19, only 7.8% were attributable to COVID-19. Two nosocomial clusters were also identified, in the emergency department (10 carers) and in the cardiology department (6 carers and one patient). However, direct diagnosis by RT-PCR has sensitivity limits and can lead to false negative results when the subject is indeed suffering from COVID-19. This lack of sensitivity is inherent to the technique on the one hand, but also to the quality of the sample and the kinetics of the infection. Indeed, the virological window during which the virus is present in the respiratory mucous membranes sampled seems relatively narrow, hence a progressive negativation of the respiratory samples as the disease progresses. Moreover, clinical symptoms vary from one individual to another, and it is now recognized that some infected persons are asymptomatic but carry the virus. Thus, the use of a second diagnostic technique is a necessity, and serology could be a relevant diagnostic support.

In the literature, several publications report the performance of COVID-19 serology in clusters of cases or cohorts of subjects. The serological techniques employed are variable (target epitopes in particular) and frequently homemade. Serology is mainly studied in comparison or association with RT-PCR in order to highlight the increased performance of COVID-19 diagnosis when the two techniques are combined. Correlation with chest CT imaging data is also encountered.

Numerous serological tests are therefore being tested to determine retrospectively whether the individual has been exposed to the virus by looking for specific antibodies to the virus. The supreme health authority has drawn up specifications dated 16 April 2020, defining the methods for evaluating the performance of serological tests detecting antibodies directed against SARSCoV-2 in order to provide a framework for these practices. Several clinical studies are also underway, in particular to assess the kinetics of the appearance of the antibodies, whether these specific antibodies would be protective and whether their appearance would coincide with a cessation of contagiousness. Thus, the main objective of this study is to evaluate the diagnostic performance of the COVID-19 immunoglobulin (IgG) Dia-Pro serological test, in view of its deployment at the Cornish Hospital Union Laboratory. Subsequently, given the low prevalence of COVID-19 in Brittany and the risk of a second epidemic wave when the confinement is lifted, the evaluation of the seroprevalence of the staff of the Cornish Hospital Union is necessary in order to assess the attack rate of COVID-19 within the establishment and particularly within departments where nosocomial clusters have been reported; and to prevent the impact of deconfinement. Indeed, knowledge of the proportion of immunized personnel and its distribution according to services will make it possible to establish internal recommendations and to effectively manage personal protective equipment inventories, in conjunction with the deconfinement strategy that will be implemented by the government. The goal is to protect hospital staff from overexposure to the virus;

ELIGIBILITY:
Inclusion Criteria:

* major
* having given his or her written consent and being able to consent
* For the prospective COVID-19 (+) sub-population : Diagnosis of COVID-19 by RT-PCR SARS-CoV-2 (+)
* For the retrospectiveCOVID-19 (+) sub-population : Serum stored as part of care in patients diagnosed with COVID-19 (+) by an RT-PCR SARS-CoV-2 (+), and no patient opposition obtained.
* For the prospective COVID-19 (-) sub-population :

No suggestive clinical picture associated with RT-PCR SARS-CoV-2 (-) or Evocative clinical picture with RT-PCR SARS-CoV-2 (-) and negative chest CT scan

* For the retrospective COVID-19 (-) sub-population : Serum kept as part of the care before the outbreak began, and no opposition from the subject obtained.
* For the staff hospital sub-population : The staff members included must be of legal age, work at the Cornish Hospital Center and have given their written consent and be able to consent.

Exclusion Criteria:

-Patients with RT-PCR SARS-CoV-2 (-) but with a chest CT suggestive of COVID-19.

And for all the patients in different sub-populations :

* incapable of consent
* refusal to participate
* not covered by a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2587 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Serological test evaluation | 1 day
  The performance of the COVID-19 IgG Dia-Pro serological test is evaluated in terms of sensitivity/specificity.

SECONDARY OUTCOMES:
Population seroprevalence | 1 month
  Population seroprevalence among hospital staff (caregivers and non-caregivers) in Quimper Hospital is assessed

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Cornouaille, Quimper, France